CLINICAL TRIAL: NCT05314374
Title: Effect of Ileocolic-released Conjugated Bile Acid on Satiety, Entero-Endocrine Cell Function, and Body Weight in Patients With Obesity and Abnormal Satiety Phenotype
Brief Title: Effect of Bile Acids on Satiety, Cell Function and Body Weight in Patients With Obesity and Abnormal Satiety Phenotype
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-008310; K23DK114460 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-04-06 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Healthy
Keywords: BMI of 30 or greater
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bile Acid Supplement Group (Experimental): Subjects with obesity and abnormal satiety phenotype will receive ileocolonic-release conjugated bile acid supplements
  Interventions: Dietary Supplement: Ileocolonic-release conjugated bile acid
- Placebo Group (Placebo Comparator): Subjects with obesity and abnormal satiety phenotype will receive matching-placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Ileocolonic-release conjugated bile acid — 500 mg tablets orally twice daily on an empty stomach, 30 minutes prior to breakfast and evening dinner for 90 +/- 5 days. Subjects will receive 500 mg twice daily during their first week and 1000 mg twice daily for the rest of the study.
  Other Names: IC-CBAS
  Arms: Bile Acid Supplement Group
Drug: Placebo — Placebo looks exactly like the study drug, but it contains no active ingredient. 500 mg tablets orally twice daily on an empty stomach, 30 minutes prior to breakfast and evening dinner for 90 +/- 5 days. Subjects will receive 500 mg twice daily during their first week and 1000 mg twice daily for the rest of the study.
  Other Names: Matching-placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to study the effect of the study drug (a conjugated bile acid dietary supplement) or placebo on cell function, hormones and body weight.

ELIGIBILITY:
Inclusion criteria:

I. Patients with obesity BMI> 30 kg/m2 and hungry gut phenotype.

II. Age: 18-65 years.

III. Gender: men or women. Women of childbearing potential will have a negative pregnancy test before initiation of medication and within 48 hours of receiving radioisotope for the gastric emptying study.

IV. Otherwise healthy individuals or with controlled chronic medical conditions such as type 2 diabetes.

Exclusion criteria:

I. Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders. For screening the bowel disease questionnaire will be used to exclude subjects with irritable bowel syndrome.

II. Subjects with stool type Bristol classification 6-7 per bowel disease questionnaire.

III. Female subjects who are pregnant or breast-feeding.

IV. Use of anti-obesity medications upon screening (ie., orlistat, phentermine-topiramate, liraglutide, semaglutide, bupropion-naltrexone), metformin or GLP-1 analogs.

V. Individuals who are currently on treatment for unstable cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine, and psychiatric disease.

VI. Any acute or chronic condition or other disease that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

VII. Significant untreated psychiatric dysfunction based upon screening. Hospital Anxiety and Depression Inventory (HAD) score >11 on depression scale, a self-administered alcoholism screening test (AUDIT-C) score >4 in men or >3 in women, and difficulties with substance or eating disorders determined by the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia); will mean the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up. The provider will review the patient's alcohol intake over the past few months to confirm accuracy and determine study eligibility.

VII. Principal Investigator discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bile Acid Supplement Group: Subjects with obesity and abnormal satiety phenotype will receive ileocolonic-release conjugated bile acid supplements
  Ileocolonic-release conjugated bile acid: 1000mg tablets orally twice a daily on an empty stomach, 30 minutes prior to breakfast and evening dinner for 90 +/- 4 days
- Placebo Group: Subjects with obesity and abnormal satiety phenotype will receive matching-placebo
  Placebo: Placebo looks exactly like the study drug, but it contains no active ingredient. 1000mg tablets orally twice a daily on an empty stomach, 30 minutes prior to breakfast and evening dinner for 90 +/- 4 days.
Period: Overall Study
Arm/Group | Bile Acid Supplement Group | Placebo Group
Started | 18 | 17
Completed | 16 | 15
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bile Acid Supplement Group | Placebo Group | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (9.7) | 49.4 (9.8) | 48.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Weight, kg [Mean (Standard Deviation); unit: kg] | 106.7 (18.5) | 108.1 (24.3) | 107 (22)
Height, m [Mean (Standard Deviation); unit: m] | 1.7 (0.1) | 1.7 (0.1) | 1.7 (0.1)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 35.3 (4) | 37.9 (5.3) | 36 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Glucagon-Like Peptide-1 (GLP-1)
Description: The number of participants that provided a blood sample for GLP-1 (ug/ml) .
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bile Acid Supplement Group | Placebo Group
Number analyzed (Participants) | 18 | 17
Participants | 18 | 17

2. Primary Outcome: Peptide Trosin Tyrosine (PYY) Hormone
Description: The number of participants that provided a blood sample for PYY.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bile Acid Supplement Group | Placebo Group
Number analyzed (Participants) | 18 | 17
Participants | 18 | 17

3. Secondary Outcome: Change in Weight
Description: Change in weight, measured in kilograms (kg), from baseline visit to 12 weeks.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Bile Acid Supplement Group | Placebo Group
Number analyzed (Participants) | 18 | 17
kg | -0.82 [-3.58 to 1.95] | 0.12 [-1.86 to 2.10]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through completion of the study, approximately 12 weeks.
Arm/Group | Bile Acid Supplement Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 14/18 | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bile Acid Supplement Group (N=18) | Placebo Group (N=17)
Diarrhea (Gastrointestinal disorders) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05314374/Prot_SAP_000.pdf